CLINICAL TRIAL: NCT00767468
Title: A Phase IB Study of Sorafenib for Patient With Locally Advanced or Metastatic Hepatocellular Carcinoma and Child's B Cirrhosis
Brief Title: Sorafenib in Treating Patients With Locally Advanced or Metastatic Liver Cancer and Cirrhosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding unavailable
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0717; P30CA016086 (NIH); CDR0000615311 (Other: PDQ number); BAYER-UNC-LCCC-0717
Record Dates: First submitted 2008-10-04; First posted 2008-10-07 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; advanced adult primary liver cancer; localized unresectable adult primary liver cancer; recurrent adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bilirubin Normal to 3x Upper Limit of Normal (Experimental)
  Interventions: Drug: sorafenib tosylate
- Bilirubin >3x to 6x Upper Limit of Normal (Experimental)
  Interventions: Drug: sorafenib tosylate

INTERVENTIONS:
Drug: sorafenib tosylate — Sorafenib 400mg BID until disease progression or patient withdrawal.
  Other Names: Sorafenib; Nexavar

SUMMARY:
RATIONALE: Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase I trial is studying the side effects and best dose of sorafenib in treating patients with locally advanced or metastatic liver cancer and cirrhosis.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the pharmacokinetic parameters of sorafenib tosylate in patients with locally advanced or metastatic hepatocellular carcinoma and Child-Pugh B cirrhosis.
* To correlate the pharmacokinetic parameters of sorfenib tosylate with hepatic retention and clearance of technetium Tc 99m mebrofenin (MEB) and technetium Tc 99m sestamibi (MIBI).

Secondary

* To establish a tolerable dose of sorafenib tosylate based on degree of liver dysfunction (bilirubin ≤ 3 times upper limit of normal [ULN] or bilirubin > 3 times but ≤ 6 times ULN).
* To correlate the pharmacokinetics MEB and MIBI with the dose-limiting toxicity of sorafenib tosylate.
* To explore whether increase in bilirubin consists primarily of conjugated or unconjugated bilirubin in response to sorafenib tosylate.
* To explore whether there is a correlation between increased bilirubin and decreased clearance of MEB and/or MIBI.
* To explore whether there is a correlation between survival and MRI characteristics associated with high tumor VEGF levels.
* To assess VEGF levels directly in available biopsy samples using IHC.
* To determine expression levels of hepatic transport proteins (i.e., OATPs, Pgp, or MRPs) that may correlate with clearance of sorafenib tosylate.
* To explore whether there is a correlation between survival and activation of the RAF/MEK/ERK pathway at baseline.
* To estimate median overall survival.

OUTLINE: This is a multicenter study. Patients are stratified according to degree of hepatic dysfunction (moderate [bilirubin ≤ 3 times upper limit of normal (ULN)] vs severe [bilirubin > 3 times but ≤ 6 times ULN]).

Patients receive oral sorafenib tosylate twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients undergo hepatic scintigraphy with technetium Tc 99m mebrofinin (MEB) and technetium Tc 99m sestamibi (MIBI) at baseline. Blood and urine samples are collected periodically for pharmacokinetic studies.

After completion of study therapy, patients are followed at 3-4 weeks and then every 3 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of hepatocellular carcinoma (HCC) according to tissue histology* NOTE: *Recurrence of previously resected HCC does not require tissue confirmation if there is clear radiographic recurrence, in the opinion of the investigator
* Locally advanced or metastatic disease OR not eligible for surgical resection or immediate liver transplantation
* Child-Pugh class B cirrhosis

  * Moderate hepatic dysfunction (bilirubin ≤ 3 times upper limit of normal [ULN]) OR severe hepatic dysfunction (bilirubin > 3 times but ≤ 6 times ULN)
* No known brain metastasis unless the metastasis has been stable for > 3 months

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy > 12 weeks
* Hemoglobin > 9.0 g/dL
* ANC > 1,000/mm^3
* Platelet count > 45,000/mm^3
* ALT and AST < 7 times ULN
* INR < 2.0
* Creatinine < 1.7 times ULN OR creatinine clearance > 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 2 weeks after completion of study treatment
* No history of uncontrolled seizures, CNS disorders, or psychiatric disability that, in the opinion of the investigator, is clinically significant, precludes giving informed consent, or interferes with compliance of oral drug intake
* No other concurrent active malignancy
* No active clinically serious infection > CTCAE grade 2
* No known hypersensitivity to sorafenib tosylate or to any of the excipients
* No known or suspected allergy to sorafenib tosylate or to any agent given in the course of this study
* No NYHA class III or IV congestive heart failure
* No unstable angina
* No new onset angina (i.e., within the past 3 months)
* No myocardial infarction within the past 6 months
* No cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* No uncontrolled hypertension, defined as systolic blood pressure (BP) > 150 mm Hg or diastolic BP > 90 mm Hg, despite optimal medical management
* No thrombolic or embolic events (e.g., cerebrovascular accident, including transient ischemic attacks) within the past 6 months
* No pulmonary hemorrhage/bleeding event > CTCAE grade 2 within the past 4 weeks
* No other hemorrhage/bleeding event > CTCAE grade 3 within the past 4 weeks
* No variceal bleeding within the past 90 days
* No known grade 2 or 3 esophageal varices
* No evidence or history of bleeding diathesis or coagulopathy
* No significant traumatic injury within the past 4 weeks
* No serious non-healing wound, ulcer, or bone fracture
* No other serious uncontrolled medical condition (e.g., uncontrolled ascites or encephalopathy) that, in the opinion of the investigator, may compromise study participation
* No condition that would impair the patient's ability to swallow whole pills
* No malabsorption problem
* No active drug or alcohol abuse

PRIOR CONCURRENT THERAPY:

* No more than one prior therapy including, but not limited to, any of the following:

  * Systemic chemotherapy
  * Hepatic artery infusion of chemotherapy
  * Chemoembolization
  * Radioembolization
  * Ablation
* At least 4 weeks since prior embolization, resection, or ablation
* No prior RAF/MEK/ERK-targeting therapy or VEGF-targeting therapy
* More than 4 weeks since prior participation in an investigational drug study
* More than 4 weeks since prior major surgery or open biopsy
* No concurrent chronic anticoagulation other than 1 mg of warfarin per day for central venous catheter patency
* No concurrent St. John's wort or rifampin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-10; Primary Completion 2010-02 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Correlation between hepatic retention and clearance of technetium Tc 99m mebrofenin (MEB) and technetium Tc 99m sestamibi (MIBI) and clearance (and other pharmacokinetic parameters) of sorafenib tosylate | 4 years

SECONDARY OUTCOMES:
Tolerable dose of sorafenib tosylate | 4 years
Correlation between the pharmacokinetics of MEB and MIBI and the dose-limiting toxicity of sorafenib tosylate | 4 years
Conjugated or unconjugated bilirubin increase in response to sorafenib tosylate | 4 years
Correlation between increased bilirubin and decreased clearance of MEB and/or MIBI | 4 years
Correlation between survival and MRI characteristics associated with high tumor VEGF levels | 4 years
Correlation between clearance of sorafenib tosylate and expression levels of hepatic transport proteins | 4 years
Correlation between survival and activation of the RAF/MEK/ERK pathway at baseline | 7 years
Median overall survival | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Bert H. O'Neil, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina